CLINICAL TRIAL: NCT05575635
Title: A Single Arm, Single Center Clinical Study of Fruquintinib Combined With Concurrent Chemoradiotherapy for Neoadjuvant Treatment of Locally Advanced Rectal Cancer
Brief Title: Neoadjuvant Treatment of Fruquintinib Combined With Concurrent Chemoradiotherapy for LARC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Ming Yue, Professor, Henan Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-C121
Record Dates: First submitted 2022-10-08; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Rectal Cancer
Keywords: neoadjuvant; peri-operative
MeSH Terms: conditions — Rectal Neoplasms | interventions — HMPL-013; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fruquintinib + mFOLFOX6 + radiotherapy (Experimental): fruquintinib + mFOLFOX6 + radiotherapy
  Interventions: Drug: fruquintinib + concurrent radiotherapy + chemotherapy

INTERVENTIONS:
Drug: fruquintinib + concurrent radiotherapy + chemotherapy — mFOLFOX6: The mFOLFOX6 regimen will be administered on Day 1 of each treatment cycle. This regimen consists of oxaliplatin 85 mg/m2 IV given over 2 hours, leucovorin 400 mg/m2 IV given over 2 hours, and fluorouracil 400 mg/m2 IV bolus, followed by fluorouracil 1200 mg/m2 per day for 2 days, continuous infusion.
  fruquintinib: 3mg/d, qd po, for 7 weeks continuously.
  Radiation Therapy: radiation 45.0~50.0 Gy (1.8-2.0 Gy/day or 25 fractions weeks 3-7)

SUMMARY:
The study aims to evaluate the efficacy and safety of fruquintinib combined with mFOLFOX6 + synchronous radiotherapy as neoadjuvant therapy in middle and low locally advanced rectal cancer patients with no previous anti-tumor treatment.

DETAILED DESCRIPTION:
The study aims to evaluate the efficacy and safety of fruquintinib combined with mFOLFOX6 + synchronous radiotherapy as neoadjuvant therapy in middle and low locally advanced rectal cancer patients with no previous anti-tumor treatment. Approximately 40 patients will be enrolled and undergo combination neoadjuvant therapy, followed by TME and mFOLFOX6 adjuvant therapy, peri-operative treatment will last for 6 months. The primary endpoint is pCR.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed rectal adenocarcinoma, classified as stage II (T3-4N0) or stage III (T1-4N1-2) by MRI and CT;
* Middle and low rectal cancer with the lower pole of the tumor less than 12 cm from the anal margin;
* The multidisciplinary cancer committee recommended neoadjuvant radiotherapy, chemotherapy and surgery;
* ECOG PS 0-1;
* Expected survival ≥ 2 years;
* Have not received any anti-tumor treatment;
* Have at least one measurable lesion;
* Sufficient organs and bone marrow functions;
* Women of childbearing age need to take effective contraceptive measures;

Exclusion Criteria:

* Patients with surgical contraindication;
* Patients with familial adenomatous polyposis (FAP), hereditary nonpolyposis colorectal cancer (HNPCC), active Crohn's disease or active ulcerative colitis;
* Other malignant tumors found within 5 years before enrollment, except skin basal cell or squamous cell carcinoma, or cervical carcinoma in situ after radical surgery;
* Serious cardiovascular disease, including unstable angina pectoris or myocardial infarction, occurred within 6 months before enrollment;
* International normalized ratio (INR)>1.5 or partially activated prothrombin time (APTT)>1.5 × ULN；
* Investigators judged clinically significant electrolyte abnormalities;
* Hypertension that could not be controlled by drugs before enrollment, which was defined as: systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg;
* Poorly controlled diabetes mellitus before enrollment (fasting glucose concentration ≥ CTCAE level 2 after regular treatment);
* Active ulcer of stomach and duodenum, ulcerative colitis and other digestive tract diseases before enrollment, or other conditions that may cause gastrointestinal bleeding and perforation judged by the researcher;
* Serious active bleeding, hemoptysis (>5 mL fresh blood within 4 weeks) or thromboembolism (including stroke and/or transient ischemic attack) occurred within 12 months before enrollment;
* Cardiovascular diseases with significant clinical significance, including but not limited to acute myocardial infarction, severe/unstable angina pectoris or coronary artery bypass grafting within 6 months before enrollment; Congestive heart failure New York Heart Association (NYHA) grade>2; Ventricular arrhythmias requiring medication; LVEF<50%;
* Active or uncontrollable serious infection (≥ CTCAE v5.0 grade 2 infection);
* Known human immunodeficiency virus (HIV) infection. A known history of liver disease with clinical significance, including viral hepatitis [People who are known to be carriers of hepatitis B virus (HBV) must exclude active HBV infection, that is, HBV DNA positive (>1 × 104 copies/mL or>2000 IU/ml); Known hepatitis C virus infection (HCV) and HCV RNA positive (>1 × 103 copies/mL);
* Unrelieved toxic reaction caused by any previous anti-cancer treatment higher than CTCAE v5.0 grade 1 or above;
* Routine urine test showed that urinary protein ≥ 2+, and 24-hour urinary protein volume>1.0g.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
pCR | about 2 months
  pathological complete response rate assessed by the investigator

SECONDARY OUTCOMES:
MPR | about 2 months
  major pathological response rate assessed by the investigator
ORR | about 2 months
  objective response rate assessed by the investigator
R0 resection rate | about 2 months
  R0 resection rate
DFS | about 3 years
  DFS (Disease-free survival) will be calculated from the date of first administration of study drug to the date of recurrence or death by any reason.
OS | about 5 years
  OS will be calculated from the date of first administration of study drug to the date of death by any reason.
TRAEs | about 6 months
  treatment-related adverse events by CTCAE v5.0